CLINICAL TRIAL: NCT04843969
Title: Investigating Stress-Potentiated Memory Updating as a Novel Intervention for Non-Treatment Seeking Smokers
Brief Title: Investigation of Cigarette Cravings in Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marco Leyton (Other)
Responsible Party: Sponsor-Investigator, Marco Leyton, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 421-0318
Record Dates: First submitted 2021-04-03; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cigarette Smoking; Addiction Nicotine; Tobacco Use
Keywords: Memory updating; Reconsolidation
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stress task and smoking cue (Experimental): Exposure to a psychosocial stress task followed by smoking video cues
  Interventions: Behavioral: Stress induction; Behavioral: Cue induction
- Stress task and neutral cue (Experimental): Exposure to a psychosocial stress task followed by neutral video cues
  Interventions: Behavioral: Stress induction; Behavioral: Neutral cue exposure
- Control task and smoking cue (Active Comparator): Exposure to a control task followed by smoking video cues
  Interventions: Behavioral: Control stress exposure; Behavioral: Cue induction
- Control task and neutral cue (Active Comparator): Exposure to a control task followed by neutral video cues
  Interventions: Behavioral: Control stress exposure; Behavioral: Neutral cue exposure

INTERVENTIONS:
Behavioral: Stress induction — Exposure to a psychosocial stressor
  Arms: Stress task and neutral cue; Stress task and smoking cue
Behavioral: Control stress exposure — Exposure to a control task (no stress)
  Arms: Control task and neutral cue; Control task and smoking cue
Behavioral: Cue induction — Exposure to a smoking-related task
  Arms: Control task and smoking cue; Stress task and smoking cue
Behavioral: Neutral cue exposure — Exposure to neutral cues
  Arms: Control task and neutral cue; Stress task and neutral cue

SUMMARY:
Interventions to disrupt memory reconsolidation have held promise for the treatment of stress- and anxiety-related disorders. In the present study, the investigators will examine whether an intervention based on these principles, called memory updating, could be adapted for reward-seeking behaviors. To test this, non-treatment seeking tobacco smokers will be exposed to smoking cues and/or stress, two stimuli known to trigger smoking. It is predicted that exposure to a stress task will enhance the cues' motivational salience and yield greater susceptibility to the memory updating procedure.

As an add-on, the investigators will examine COVID-associated changes in substance use and whether participants in the memory updating groups might be more resilient to these effects. It is predicted that the changes in substance use will depend on whether the substances are used primarily in social settings.

DETAILED DESCRIPTION:
Non-treatment seeking cigarette dependent smokers will be randomized to one of four testing conditions: 1) a non-stressful task followed by neutral cues, 2) the non-stressful task followed by smoking cues, 3) a stressful task followed by neutral cues, or 4) the stressful task followed by smoking cues. Ten minutes after the intervention, participants will undergo a 60-minute extinction procedure consisting of smoking-related videos, images and smoking paraphernalia. Cue reactivity test sessions will take place 24 hours, 2 weeks and 6 weeks following the intervention.

COVID-associated changes in substance use will be quantified over three telephone interviews: one at the end of March / beginning of April 2020 (at the start of the pandemic), one at the end of April / beginning of May, and a final one which will be instituted if feasible once the infection rates and social distancing policies have decreased.

ELIGIBILITY:
Inclusion Criteria:

* Scoring 5 or higher on the Fagerström Test for Cigarette Dependence
* Willingness to abstain from smoking for 4 hours prior to each laboratory visit

Exclusion Criteria:

* Currently using cigarette cessation products
* Endocrinological problems
* Significant mental or physical health conditions
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in cigarettes smoked per day from the pre-intervention baseline to test sessions 2 and 3 given two and six weeks post-intervention | At the end of test session 1 (24 hours post-intervention), participants will receive a journal to record their daily smoking behaviour. They are asked to keep this journal until test session 3 (6 weeks post-intervention).
  A journal is given to participants to record their cigarette use behaviour every day for a month and a half

SECONDARY OUTCOMES:
Change in smoking cue-induced cigarette cravings from the pre-intervention baseline to test session 2 | Multiple times points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention.
  Participants will be asked to complete craving and urge to smoke questionnaires at several time points throughout the study sessions
Change in smoking cue-induced cigarette cravings from the pre-intervention baseline to test session 3 | Multiple times points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention.
  Participants will be asked to complete craving and urge to smoke questionnaires at several time points throughout the study sessions
Change in smoking cue-induced heart rate responses from the pre-intervention baseline to test session 2 | Multiple time points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention
  Participants' heart rate will be measured through the use of a polar belt at several time points during the study sessions
Change in smoking cue-induced heart rate responses from the pre-intervention baseline to test session 3 | Multiple time points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention
  Participants' heart rate will be measured through the use of a polar belt at several time points during the study sessions
Change in smoking cue-induced skin conductance responses from the pre-intervention baseline to test session 2 | Multiple time points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention
  Participants' skin conductance will be measured through the use of electrodes on their index and middle fingers at several time points during the study sessions
Change in smoking cue-induced skin conductance responses from the pre-intervention baseline to test session 3 | Multiple time points during the baseline, intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention
  Participants' skin conductance will be measured through the use of electrodes on their index and middle fingers at several time points during the study sessions
Change in tobacco and other substance use patterns from the pre-COVID-19 baseline to during COVID-19 | Multiple time points at baseline (before the pandemic), at the start of the pandemic, and during the pandemic
  Participants will be asked to report the quantity of cigarettes and/or other substances they have consumed recently
Change in tobacco and other substance use patterns from the pre-COVID-19 baseline to post-COVID-19 | At baseline (before the pandemic) and through study completion, an average of 1 year
  Participants will be asked to report the quantity of cigarettes and/or other substances they have consumed recently
Change in tobacco and other substance use patterns during the COVID-19 pandemic to post-COVID-19 | Multiple time points during the pandemic and through study completion, an average of 1 year
  Participants will be asked to report the quantity of cigarettes and/or other substances they have consumed recently

OTHER OUTCOMES:
Change in stress- and/or cue-induced mood during the intervention and at test sessions 1, 2 and 3 | Multiple time points during the intervention and test sessions at 24 hours, 2 weeks and 6 weeks post-intervention
  Participants will be asked to complete a mood questionnaire at several time points during the intervention and at test sessions 1, 2 and 3
Change in cigarette use over the course of the procedure as a function of personality factors, childhood trauma, perceived stress, mood and/or cigarette withdrawal | Multiple time points at baseline, during the intervention, at test sessions (24 hours, 2 weeks and 6 weeks post-intervention) and telephone follow-ups (6 months post-intervention)
  Participants will be asked to complete self-report questionnaires about their personality traits, traumatic childhood experiences, perceived stress, current mood states and cigarette withdrawal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Marco Leyton, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified individual participant data that underlie any results reported in the article. This includes results reported in text, figures and appendices.
Time Frame: From 9 to 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has already been approved by an ethics committee.

REFERENCES:
- [Derived] Barnabe A, Gamache K, de Camargo JVP, Allen-Flanagan E, Rioux M, Pruessner J, Leyton M, Nader K. A novel stress-based intervention reduces cigarette use in non-treatment seeking smokers. Neuropsychopharmacology. 2023 Jan;48(2):308-316. doi: 10.1038/s41386-022-01455-6. Epub 2022 Sep 29. PMID 36175551